CLINICAL TRIAL: NCT04259866
Title: FALSE POSITIVE FINDINGS IN BREAST CANCER TOMOSYNTHESIS: An Analysis of Findings Leading to Recall and Work-up in ASL Avellino Screening
Brief Title: FALSE POSITIVE FINDINGS IN BREAST CANCER TOMOSYNTHESIS
Status: Completed | Type: Observational
Sponsor: "G Criscuoli" Hospital (Other)
Responsible Party: Principal Investigator, Graziella Di Grezia, 1st level Assistant Physician, Azienda Sanitaria ASL Avellino 2
Other Study IDs: 05022020
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To analyse false positives in breast cancer screening with tomosynthesis versus 2D mammography. The Avellino Breast Tomosynthesis Screening Trial is a observational population-based study that analyze souspicious findings in tomosynthesis slice images.

This study is based on two years screening and tomosynthesis was analzyed by two expert breast radiologists.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer screening population

Exclusion Criteria:

* previous cancer
* breast prostheses

Ages: 50 Years to 69 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: female population candidated to breast cancer screening program
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
recall rate | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Graziella Di Grezia, Avellino, Av, Italy

IPD SHARING:
Plan to Share IPD: Undecided